CLINICAL TRIAL: NCT02302651
Title: Treatment of Osteoid Osteoma With MR Guided High Intensity Focused Ultrasound
Brief Title: Non-invasive Focal Therapy for Osteoid Osteoma
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Alessandro Napoli, MD, PhD, University of Roma La Sapienza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OO-MC-MRGFUS-002
Record Dates: First submitted 2014-11-19; First posted 2014-11-27 (Estimated); Last update posted 2014-11-27 (Estimated); Status verified 2014-11

CONDITIONS: Osteoma, Osteoid
Keywords: high intensity focused ultrasound; osteoid osteoma; bone tumor
MeSH Terms: conditions — Osteoma, Osteoid; Bone Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Osteoid Osteoma (Other): MR guided High Intensity focused ultrasound
  Interventions: Device: MR guided High Intensity focused ultrasound

INTERVENTIONS:
Device: MR guided High Intensity focused ultrasound — High Intensity Focused Ultrasound is a totally non-invasive procedure that can destroy tumors transcutaneously; safety and efficacy profile are dramatically increased by the MRI guidance

SUMMARY:
Non-invasive treatment of Osteoid osteoma using MRI guided high-intensity focused ultrasound. This study is designed as an intention-to-treat using a totally non-invasive approach for pain reduction, quality of life improvement and long-term bone restoration. Procedure is performed in a single session using limited amount of acoustic energy to target the osteoid nidus. Treatment will be performed under anesthesia (peripheral or general according to age and lesion position).

DETAILED DESCRIPTION:
An osteoid osteoma is a benign, painful musculoskeletal tumor that usually occurs in young males. The standard of care in the United States is computed tomography (CT)-guided radiofrequency ablation, a minimally invasive percutaneous procedure, with clinical success rates ranging between 85% and 98%.

Percutaneous or surgical therapy can lead to non-negligible side-effects and limited efficacy for pediatric population or young adults with osteoid osteoma. We investigate whether selective focal ablation of osteoid lesions can reduce this treatment burden without compromising long-term clinical efficacy.

Treatments will be performed using a 3.0-T MR unit (Discovery MR 750; GE Medical Systems, Milwaukee,Wis) featuring a Conformité Européenne-approved ExAblate MR-guided focused ultrasound system (InSightec,Tirat-Carmel, Israel) in which the ultrasound transducer is housed in the patient table. Alignment between the lesion and the transducer will be obtained in each patient by using a moistened gel pad and degassed water for acoustic coupling. This approach avoided air- skin interfaces, which can cause energy reflection and skin burns. After patient positioning, the lesion is localized with MR for treatment by using variably orientated non enhanced T1- and T2-weighted acquisitions. In general, an ideal 90° incidental angle between the planned focused ultrasound path and the lesion, relative to the bone long axis, is obtained or at least approximated. The shortest skin-lesion distance is selected for the beam pathway. Care will be taken to avoid multiple interfaces (skin, muscle, fasciae) as much as possible so as to minimize deflection of the focused ultrasound beam. Each lesion will be manually segmented by the operator to precisely delineate the nidus, skin surface, and cortical surface of the bone. Sensitive areas surrounding the target volumes will also be drawn to limit the energy and prevent unwanted thermal damage. The treatment plan is than calculated automatically by the ExAblate software according to previously acquired parameters, including the energy (in joules), the interval between two sonications, the sonication duration, and the spot size, which are modifiable by the operator. Thereafter, a low-energy sonication test will be performed to confirm the path and correct direction of the ultrasound beam into the target area and to confirm the planned energy dose and the effective dose deployed to the lesion.

The increase in tissue temperature is evaluated by using real-time MR thermometry of phase-difference fast spoiled gradient-echo sequences (proton resonant frequency shift method). The sequences are acquired to provide temperature-dependent images and real-time mapping of the thermal dose on a preferred imaging plane. The proton resonant frequency shift method starts simultaneously with each sonication. Similar to other treatments of bone lesions that use MR-guided focused ultrasound, the temperature increase is determined on the adjacent periskeletal tissue. In fact, proton resonant frequency sequences cannot effectively measure the temperature on the bone surface because of the absence of moving protons in the cortical zone. Thus, MR thermometry reveals a temperature increase, which propagates by conductive processes from the bone to the immediately adjacent soft tissues that respond linearly to an increase in bone temperature, thereby allowing an accurate measure of heating. Portions of periosteum and adjacent tumor that are not fully ablated can be re-treated if deemed necessary. The critical temperature threshold for ablation is set at 65°C in the soft tissues adjacent to the targeted bone structures. Postprocedural care includes evaluation of possible skin burns, monitoring of vital signs for 2 hours after treatment in the MR department, and administration of analgesic and/or antiemetic drugs if requested. Treatment-related adverse events will be recorded as minor or major on the basis of medical severity, additional treatment, and long-term consequences for patients. Treatment will be performed on an outpatient basis in the patients who receive only local and peripheral anesthesia; the patient who receives general anesthesia is usually hospitalized for 24 hours after treatment.

ELIGIBILITY:
Inclusion Criteria:

* clinical and imaging diagnosis of osteoid osteoma
* painful non-vertebral location

Exclusion Criteria:

* general contraindication to MRI
* vertebral location of the lesion
* claustrophobia and prior surgery or RFA are not an absolute exclusion criterion

Ages: 3 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-06; Primary Completion 2015-06 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Safety - Adverse Events (serious and otherwise) | 1 year
  to assess complications
Efficacy (Symptoms reduction) | 4 years
  Symptoms reduction

SECONDARY OUTCOMES:
nidus vascularization (correlation between nidus vascularization reduction and symptoms relieve) | 4 years
  correlation between nidus vascularization reduction and symptoms relieve

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro napoli, MD, PhD, Principal Investigator — Sapienza University of Rome, Policlinico Umberto I Hospital
Locations (1):
- Alessandro Napoli, Rome, Italy

REFERENCES:
- [Derived] Napoli A, Bazzocchi A, Scipione R, Anzidei M, Saba L, Ghanouni P, Cozzi DA, Catalano C. Noninvasive Therapy for Osteoid Osteoma: A Prospective Developmental Study with MR Imaging-guided High-Intensity Focused Ultrasound. Radiology. 2017 Oct;285(1):186-196. doi: 10.1148/radiol.2017162680. Epub 2017 Jun 7. PMID 28590796